CLINICAL TRIAL: NCT00808145
Title: A Phase II Study of Sorafenib With Gemcitabine/Cisplatin in Advanced Hepatocellular Carcinoma
Brief Title: Study of Sorafenib, Gemcitabine, and Cisplatin in Advanced Hepatocellular Carcinoma (HCC)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment, many screen failures and non eligible study participants
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-108
Record Dates: First submitted 2008-12-11; First posted 2008-12-15 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: Treatment of advanced liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Gemcitabine; Cisplatin; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine/Cisiplatin/Sorafenib (Experimental): All eligible patients will receive intravenous gemcitabine/cisplatin + daily oral sorafenib until disease progression occurs
  Interventions: Drug: Gemcitabine / Cisplatin / Sorafenib

INTERVENTIONS:
Drug: Gemcitabine / Cisplatin / Sorafenib — All patients will receive gemcitabine 1000mg/m2 cisplatin 30mg/m2 sorafenib 400mg orally twice daily
  Other Names: nexavar - sorafenib; gemzar - gemcitabine; cisplatin

SUMMARY:
This study will look at the safety and efficacy of treating advanced hepatocellular carcinoma in patients who have not yet received systemic chemotherapy. Previous local treatment of hepatic lesions is permitted The treatment will use a combination of three FDA approved chemotherapy drugs, Gemcitabine, Cisplatin and Sorafenib. Sorafenib is FDA approved for the treatment of hepatocellular cancer, gemcitabine and cisplatin are not approved for the treatment of hepatocellular cancer.

DETAILED DESCRIPTION:
This study will look at the effectiveness and safety of combining gemcitabine, cisplatin and sorafenib for the treatment of advanced hepatocellular carcinoma in patients with advanced disease who are chemo naive. Sorafenib has shown an increase in median survival but only tumor shrinkage by RECIST criteria. Since much of the morbidity and mortality of this disease occurs due to continued tumor growth in an already compromised liver, decreasing the size of the tumors might have significant impact on survival. The addition of traditional cytoxic agents might cause measureable tumor response and add to the survival benefit already seen with sorafenib. Gemcitabine and cisplatin are agents commonly used for systemic treatment of this disease and have demonstrated some effectiveness in disease control rate and median time to progression. Gemcitabine/Cisplatin have been used safely in combination with sorafenib in patients with lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma: diagnosed histologically, cytologically, or clinically by a rising AFP > 500 ng/ml in the setting of cirrhosis and a radiographically compatible lesion.
* No prior systemic therapy; local therapy such as chemoembolization, radiofrequency ablation or cryoablation is allowed.
* Measurable disease > 1 cm by CT or MRI. Lesions which have received local therapy do not qualify as measurable target lesions.
* Age > 18 years old
* ECOG Performance Status 0 or 1
* Child-Pugh status A and B
* Adequate bone marrow, liver and renal function as assessed by the following:

  * Hemoglobin ≥ 9.0 g/dl
  * Absolute neutrophil count (ANC) ≥ 1,250/mm3
  * Platelet count ≥ 80,000/mm3
  * Total bilirubin ≤ 3.0 mg/dl
  * ALT and AST ≤ 5 times the ULN
  * Amylase and lipase ≤ 1.5 times ULN
  * Creatinine ≤ 1.5 times ULN
* Resolution of all acute toxic effects of any prior local treatment to CTC Adverse Events grade £1.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Men should use adequate birth control for at least three months after the last administration of sorafenib.
* Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.
* INR < 1.5 or a PT/PTT within normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the INR or PT and PTT should be measured prior to initiation of sorafenib and monitored at Day 1 and Day 8 of each cycle.

Exclusion Criteria:

* Prior surgery, radiation or local therapy within 4 weeks.
* Prior treatment with either sorafenib, gemcitabine, or cisplatin
* Cardiac disease: Congestive heart failure > class II NYHA. Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* Known brain metastasis. Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension defined as sustained systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
* Known human immunodeficiency virus (HIV) infection
* Active clinically serious infection > CTCAE Grade 2.
* Thrombotic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Serious non-healing wound, ulcer, or bone fracture.
* Evidence or history of bleeding diathesis or coagulopathy
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
* Use of St. John's Wort or rifampin (rifampicin).
* Known or suspected allergy to sorafenib, cisplatin, or gemcitabine.
* Any condition that impairs patient's ability to swallow whole pills.
* Any malabsorption problem.
* Uncontrolled ascites (defined as not easily controlled with diuretic treatment).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Safety of the combination of gemcitabine/cisplatin/sorafenib | one year

SECONDARY OUTCOMES:
Effectiveness of gemcitabine/cisplatin/sorafenib in shrinking tumors extending time to progression of disease | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Keith E. Stuart, M.D., Principal Investigator — Lahey Clinic
Locations (1):
- Lahey Clinic, Burlington, Massachusetts, United States